CLINICAL TRIAL: NCT02960659
Title: Therapeutic Targets in African-American Youth With Type 2 Diabetes
Brief Title: Title: Therapeutic Targets in African-American Youth With Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 170013; 17-DK-0013 (Other: NIH Clinical Center)
Record Dates: First submitted 2016-11-09; First posted 2016-11-10 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-04-12

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Metformin; Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Liraglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): Standard release metformin (500 mg tablets) was initiated and titrated to maximum dose of metformin 1000 mg twice daily over 3 weeks and continued for 12 weeks
  Interventions: Drug: Metformin
- Metformin and liraglutide (Experimental): Standard release metformin (500 mg tablets) and liraglutide (0.6mg) were initiated and titrated to maximum dose of metformin 1000 mg twice daily, and liraglutide 1.8 mg daily over 3 weeks and continued for 12 weeks
  Interventions: Drug: Liraglutide; Drug: Metformin

INTERVENTIONS:
Drug: Liraglutide — Liraglutide (6mg/ml, 3ml ) solution for subcutaneous injection, pre-filled, multi-dose pen that delivers doses of 0.6mg, 1.2mg or 1.8mg.
  Arms: Metformin and liraglutide
Drug: Metformin — Metformin 500mg oral tablet

SUMMARY:
Background:

The pill metformin treats diabetes. But it does not work for all youth, especially African-Americans. The injectable Liraglutide treats type 2 diabetes in adults. Researchers want to understand how these drugs work and if they decrease excess sugar made by the liver in youth with type 2 diabetes.

Objective:

To test if using liraglutide and metformin are better than just metformin for decreasing excess sugar produced by the liver in African-American youth with type 2 diabetes.

Eligibility:

African-Americans ages 12-25 with type 2 diabetes

Design:

Visit 1: Participants will be screened with medical history, physical exam, and blood and urine tests. Participants will stop taking diabetes medicines for 1 week. They will learn how to check blood sugars at home twice a day.

Visit 2: Overnight at the clinic. Participants will have:

Vital signs taken.

Pregnancy test.

A thin plastic tube (IV catheter) be inserted in each forearm by needle.

Blood drawn several times after drinking a sweet drink.

X-ray of total body fat.

Urine and stool collected.

Breath tests while wearing a clear hood for up to 45 minutes.

For several hours, participants can have only water. At 4 a.m. they will get sugar and fat with nonradioactive isotopes in one IV. Blood will be collected. Every 30 minutes from 9 a.m. to 2 p.m., they will drink small amounts of a shake and have blood drawn.

Participants will be randomly assigned to take either both study drugs daily or just metformin daily.

Visits 3-4: Participants will bring their blood sugar records and have blood tests.

Visit 5, after 3 months: Repeat of visit 2....

DETAILED DESCRIPTION:
Type 2 Diabetes in youth is an emerging public health concern that disproportionately affects minority children. Among minority youth, African-Americans have the highest complication rates, yet the reasons underlying this health disparity are not fully understood. Furthermore, current treatment options are limited, and African-American youth have high treatment failure rates. Metformin therapy is the only oral diabetes drug approved for use in youth with type 2 diabetes. However, metformin works less than 50% of the time in African-American youth and there is marked variability among individuals. Improving outcomes in youth requires understanding the way that drugs such as metformin work in youth and why it does not work in some individuals. New evidence suggests that the ability of metformin to work effectively may be influenced by certain genes or differences in gut bacteria. However, little is known about how genes or gut bacteria may affect youth, especially African-Americans.

To treat this aggressive disease, it is also necessary to simultaneously evaluate new therapeutic options, such as combination therapy of metformin with liraglutide in youth at highest risk for complications. Liraglutide is approved to treat type 2 diabetes in patient 10 years and older as an adjunct to diet and exercise. Liraglutide may be a useful early treatment in youth with type 2 diabetes because it may decrease glucose produced by the liver (an early prominent feature of type 2 diabetes in youth). This study is designed to examine the mechanism of action in the liver of these 2 agents and explore how genetic and gut factors may influence this action.

The primary objective of this pilot study is to compare the ability of two anti-diabetic regimens (metformin and liraglutide versus metformin alone) to lower gluconeogenesis (glucose produced by the liver) in African-American youth with type 2 diabetes. The secondary objectives are to evaluate the effect of these regimens on the following: (1) hepatic glucose production, and insulin sensitivity and (2) insulin and gut hormones concentrations (e.g. incretins). In addition, we will examine the relationship of known differences in genes associated with metformin transport and action with changes in gluconeogenesis and begin to explore the role of gut bacteria to metformin s glucose-lowering effect.

The study design is a parallel-randomized intervention trial of African-American youth with type 2 diabetes who are not on insulin therapy and who are within 5 years of diagnosis. Patients aged 12- 25 years with type 2 diabetes will be enrolled. Participants will be randomized into two intervention arms (16 in each group): metformin and liraglutide versus metformin alone. The study will consist of 5 visits. At Visit 1, a medical history, physical examination and screening labs will be done. Then the eligible participants will undergo a one-week drug-free run-in. At Visit 2 there will be an overnight inpatient stay to perform metabolic testing prior to starting the study drug(s). Participants will start the study drug(s) immediately after Visit 2 and remain on the study drug(s) for 12 weeks. Follow-up monitoring will be performed at 4-week intervals (Visit 3 and 4). The final visit (Visit 5) will occur after 12 weeks.

The ultimate goal of this multi-site project is to begin to address diabetes disparities in African-American youth by understanding the mechanism of action of these diabetes agents to inform precision medicine initiatives. This project brings together the skills and expertise of investigators within the National Institute of Diabetes and Digestive Disorders and Kidney Diseases (NIDDK), the National Human Genome Research Institute (NHGRI), and the Children s National Medical Center (CNMC). Patient recruitment and data collection will occur at NIH Clinical Center. Eligible patients may be identified through CNMC but no enrollment, informed consent or study visits will occur at CNMC.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Youth must self-identify as African-American and identify both parents as African-American
  2. Age 12-25 years
  3. Pubertal or post-pubertal: Girls Tanner stage IV-V breast; Boys Testicular volume 11-25cc
  4. Diagnosis of type 2 diabetes of less than or equal to 5 years duration, as per American Diabetes Association Criteria
  5. Hemoglobin A1C <9% at study initiation
  6. Negative to mild ketonuria without acidosis (negative or 1+ ketones on urinalysis)
  7. Negative test for diabetes-related autoantibodies (glutamic acid decarboxylase 65 and tyrosine phosphatase-related islet antigen 2 (IA-2))
  8. Willing and able to take daily medications and check blood glucose levels at least twice per day or wear a continuous glucose monitoring device (CGM).

EXCLUSION CRITERIA:

1. Pregnancy or breastfeeding
2. Allergy to study medications
3. Allergy to milk protein
4. Chronic insulin therapy
5. Treatment with other medications which are known to affect the parameters under study (for example sodium glucose transporter 2 (SGLT-2) inhibitors, dipeptidyl peptidase-4 (DPP-IV) inhibitors, non-selective beta blockers).
6. Metabolic derangement such as metabolic acidosis, severe hyperglycemia (fasting blood glucose greater than or equal to 200mg/dL), and/or liver enzymes > three times the upper limit of normal.
7. Personal or family history of medullary thyroid cancer or Multiple Endocrine Neoplasia syndrome type 2
8. Any other condition that, in the opinion of the investigators, will increase risk to the subject, or impede the accurate collection of study-related data.
9. Body weight greater than or equal to 450 lbs
10. Body weight less than or equal to 58kg
11. Serum triglyceride concentrations greater than or equal to 500mg/dl
12. Hemoglobin concentration <10g/dL

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Chung, MBBS, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators should contact the PI for information about data sharing

REFERENCES:
- [Derived] Glaros SB, Mishra SP, Jain S, Davis FS, Gabel SA, Mueller GA, Jarmusch AK, Mabundo L, Courville AB, Walter MF, Walter PJ, Overdahl KE, Yadav H, Chung ST. Systemic and gut microbiome changes with metformin and liraglutide in youth-onset type 2 diabetes: the MIGHTY study. Gut Microbes. 2025 Dec;17(1):2558071. doi: 10.1080/19490976.2025.2558071. Epub 2025 Sep 29. PMID 41020378
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-DK-0013.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin | Metformin and Liraglutide
Started | 13 | 11
Completed | 12 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Poor compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Metformin and Liraglutide | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.6 (2.1) | 15.0 (2.1) | 15.3 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 41.6 (7.3) | 38.2 (8.0) | 40.0 (7.7)
Absolute gluconeogenesis [Mean (Standard Deviation); unit: mg/kg LBM/min] — Population: This measurement is not available for two participant who withdrew and for one additional participant in the combination group due to technical difficulties
  mg/kg LBM/min
    number analyzed (Participants) | 11 | 10 | 21
    (all) | 1.86 (0.34) | 1.75 (0.36) | 1.81 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Change in Absolute Gluconeogenesis From Baseline to 12 Weeks
Description: Gluconeogenesis is measured using stable isotope tracers and is reported as mg/kg lean body mass (LBM) per minute
Time Frame: Baseline to 12 weeks
Population: Data are missing for one patient in the Metformin group due to technical difficulties
Measure: Mean (Standard Deviation); unit: mg/kg LBM/min
Arm/Group | Metformin | Metformin and Liraglutide
Number analyzed (Participants) | 11 | 10
mg/kg LBM/min | 0.018 (0.34) | -0.050 (0.24)

2. Secondary Outcome: Change in Glucose Production Rate From Baseline to 12 Weeks
Description: Glucose production rate is measured using stable isotope tracers and is reported as mg/kg LBM per minute.
Time Frame: Baseline to 12 weeks
Population: Data are missing for one patient in the Metformin group due to technical difficulties
Measure: Mean (Standard Deviation); unit: mg/kg LBM/min
Arm/Group | Metformin | Metformin and Liraglutide
Number analyzed (Participants) | 11 | 10
mg/kg LBM/min | 0.089 (0.28) | -0.101 (0.24)

3. Secondary Outcome: Change in GIP AUC During OGTT and Meal Absorption
Description: Change in glucose-dependent insulinotropic polypeptide (GIP) AUC during OGTT and meal absorption
Time Frame: Baseline to 12 weeks
Population: Data are missing for 3 patients in the Metformin group due to technical difficulties
Measure: Mean (Standard Deviation); unit: pg*ml/min
Arm/Group | Metformin | Metformin and Liraglutide
Number analyzed (Participants) | 9 | 10
pg*ml/min | -4432 (10550) | -1476 (11798)

4. Secondary Outcome: Change in GLP-1 Area Under the Curve Concentrations (AUC) During OGTT and Meal Absorption
Description: Change in Glucagon-like peptide-1 (GLP-1) area under the curve concentrations (AUC) during OGTT and meal absorption. These data cannot be reported at this time due to problems with the assay. It is expected that a new assay will be available by May 2024
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted, anticipated posting 2024-05

5. Secondary Outcome: Change in Whole Body Insulin Sensitivity From Baseline to 12 Weeks
Description: Whole body insulin sensitivity is estimated from a model of glucose and insulin values obtained during the OGTT and is measured in 10^-4 mU/ml/min
Time Frame: Baseline to 12 weeks
Population: Data are missing for 3 patients in the Metformin group due to technical difficulties
Measure: Mean (Standard Deviation); unit: 10^-4 mU/ml/min
Arm/Group | Metformin | Metformin and Liraglutide
Number analyzed (Participants) | 9 | 10
10^-4 mU/ml/min | 0.023 (0.045) | 0.020 (0.106)

6. Secondary Outcome: Change in Hepatic Insulin Sensitivity Index From Baseline to 12 Weeks
Description: The Hepatic Insulin Sensitivity Index(HISI) is the reciprocal of glucose rate of appearance [1000/(μmol/min)] X insulin concentration [mU/L]
Time Frame: Baseline to 12 weeks
Population: Data are missing for one patient in the Metformin group due to technical difficulties
Measure: Mean (Standard Deviation); unit: 1000mU/L/(μmol/min)
Arm/Group | Metformin | Metformin and Liraglutide
Number analyzed (Participants) | 11 | 10
1000mU/L/(μmol/min) | 0.86 (1.50) | 0.46 (1.42)

7. Secondary Outcome: Change in Insulin AUC Concentrations During an OGTT and Meal Absorption
Description: Change in insulin AUC as derived from 2-hour oral glucose tolerance test (OGTT). AUC is calculated using a trapezoidal rule. Higher AUC indicates higher insulin secretion
Time Frame: Baseline to 12 weeks
Population: Data are missing for 3 patients in the Metformin group and one patient in the combination group due to technical difficulties
Measure: Mean (Standard Deviation); unit: min*pmol/L
Arm/Group | Metformin | Metformin and Liraglutide
Number analyzed (Participants) | 9 | 9
min*pmol/L | -6381 (40108) | 47831 (48143)

8. Secondary Outcome: Change in Glycerol Turnover From Baseline to 12 Weeks
Description: Glycerol turnover is measured using stable isotope tracers and is reported as mg/kg LBM per minute.
Time Frame: Baseline to 12 weeks
Population: Data are missing for 5 patients in the Metformin group and 5 patients in the combination group due to technical difficulties
Measure: Mean (Standard Deviation); unit: mg/kg LBM/min
Arm/Group | Metformin | Metformin and Liraglutide
Number analyzed (Participants) | 7 | 5
mg/kg LBM/min | -0.057 (0.131) | -0.030 (0.104)

9. Secondary Outcome: Change in Palmitate Turnover From Baseline to 12 Weeks
Description: Palmitate turnover is measured using stable isotope tracers and is reported as mg/kg LBM per minute.
Time Frame: Baseline to 12 weeks
Population: Data are missing for 7 patients in the Metformin group and 5 patients in the combination group due to technical difficulties
Measure: Mean (Standard Deviation); unit: mg/kg LBM/min
Arm/Group | Metformin | Metformin and Liraglutide
Number analyzed (Participants) | 5 | 5
mg/kg LBM/min | 0.003 (0.24) | -0.18 (0.21)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Metformin | Metformin and Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 6/13 | 7/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=13) | Metformin and Liraglutide (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02960659/Prot_SAP_000.pdf